CLINICAL TRIAL: NCT07048795
Title: Impact de l'Utilisation du système Mylife CamAPS FX associé au Capteur DEXCOM G6 Sur le contrôle glycémique et la qualité de Vie de Patients DT1, en Vie réelle, en France
Brief Title: Impact of the Mylife CamAPS FX System With the DEXCOM G6 Sensor on T1D Patients in France
Acronym: EPICAM-G6
Status: Recruiting | Type: Observational
Sponsor: mylife Diabetes Care AG (Industry)
Collaborators: Qualees SAS (Unknown); CamDiab Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-A00207-40
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Type 1
Keywords: Diabetes Mellitus, Type 1; Hybrid closed loop system; Glycemic control; Real-life use; Semi-closed loop; Artificial pancreas; Quality of life; mylife CamAPS FX; YpsoPump; Hybrid closed loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with type 1 diabetes initiating the hybrid closed-loop system studied: Participants (adults and minors) with type 1 diabetes (T1D) initiating the mylife CamAPS FX system combined with the Dexcom G6 sensor, under real-life management conditions
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention

SUMMARY:
This is a non-interventional, longitudinal, prospective, multicenter, post market-registration and national study conducted in France. The study is conducted among participants with type 1 diabetes (T1D) using the mylife CamAPS FX hybrid closed-loop insulin delivery system combined with the DEXCOM G6 Continuous Glucose Monitoring (CGM) sensor (the System).

The main objective of the study is to evaluate, under real-life conditions, the impact of the System on glycemic control in participants with T1D after one year of use.

Secondary objectives include assessing participant-reported outcomes, such as quality-of-life, treatment satisfaction, fear of hypoglycemia, and sleep quality, describing complications related to the system, the rate of hybrid closed-loop usage over one year, and analyzing system usage parameters (e.g., Boost/Ease-Off mode use, insulin-to-carbohydrate ratios, alarms, meal announcements).

The study will involve approximately 125 participants (including 100 adults and 25 minors) across 20 centers in France.

The study is "non-interventional", which means that care and treatment are carried out as per the routine standard treatment by the endocrinologists / diabetes specialists. The decision to initiate treatment with the System is made independently of the study participation.

Participants in the study will be followed up as part of routine care at 3 visits coinciding with the three data collection time points in the study: at inclusion (baseline, Visit 0), at around 3 months (Visit 1), and around 12 months (Visit 2) after activation of the hybrid closed-loop mode.

Endocrinologists / diabetes specialists will monitor participants over the 12-month period after they start using the system and collect data at the three data collection time points. Continuous glucose sensor (CGM) and insulin pump data will also be collected.

Participants will also be asked at the three data collection time points to complete online questionnaires on their experience with diabetes.

DETAILED DESCRIPTION:
This study, called EPICAM-PMCF-G6, is part of a Post-Market Clinical Follow-up (PMCF) requested by the French Health Technology Assessment Committee (CNEDiMTS), following the listing of the System for reimbursement under the national healthcare system in France.

This study is carried following the European Regulation (EU) 2017/745 on medical devices (Medical Devices Regulation, MDR) and thus falls into the category of clinical investigations (CI) of Medical Devices (MD).

The System evaluated in this clinical investigation bears CE-marking (market approval according to the MDR) and is used in accordance with its intended purpose. As this study does not involve any invasive or burdensome procedures, it is classified as a non-invasive PMCF investigation of category 4.1. according to the French National Agency for the Safety of Medicines and Health Products (ANSM).

ELIGIBILITY:
Inclusion Criteria:

* Patient with Type 1 Diabetes using the mylife Ypsopump and the Dexcom G6 CGM sensor for at least 14 days prior to the V0 visit.
* Patient having used continuous glucose measurement with the Dexcom G6 CGM sensor at least 70% of the time during the 14-day period prior to the V0 visit.
* Patient for whom the diabetes specialist decides to initiate the mylife CamAPS FX hybrid closed loop in accordance with the reimbursement criteria applicable at the time of inclusion in the study.
* Patient who received the information sheets and gave their consent to participate in the study and to the processing of their personal data.
* Adult patient who signed an informed consent form to participate in the study or minor patient whose parents signed an informed consent form for their child's participation in the study.
* Adult patient, minor patient old enough to complete the questionnaires or parent of a minor patient able to read and understand French.
* Adult patient / minor patient capable to complete the questionnaires or parent of a minor patient who agrees to complete the online self-questionnaires.

Exclusion Criteria:

* Patient who used a hybrid closed-loop system, a fully closed-loop system, or a do-it-yourself loop system, regardless of the brand or model, within the past 6 months.
* Patient taking part or having taken part in the previous month in a diabetes trial.
* Patient or parent unable to give consent.
* Protected Patient (subject to a legal protection measure: guardianship, curatorship or legal safeguard).
* Patient with a contraindication to the prescription of the mylife CamAPS FX hybrid closed-loop ( according to the Instructions For Use, IFU).
* Patient with an unresolved skin condition in the area of sensor placement and/or in the tubing placement area (e.g. psoriasis, dermatitis herpetiformis, rash, staphylococcal infection).
* Patient with unstable diabetic retinopathy requiring laser treatment.
* Patient with associated pathology or treatment that alters glucose metabolism.
* Patient whose follow-up cannot be carried out by the centre (relocation planned within 12 months of inclusion).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be recruited from 20 French participating centers, which are defined as insulin pump initiation hospital centers according to the definition of the Francophone Diabetic Society.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Time in Range (TIR) from inclusion to 3 months | Inclusion and 3 months
  Change in Time in Range (TIR, 70-180 mg/dL; for pregnant women: TIR, 63-140 mg/dL) (%), from inclusion (hybrid closed-loop initiation) to 3 months. TIR data will be collected from system records over the 14-day period preceding each visit (inclusion and 3-month Follow-up).

SECONDARY OUTCOMES:
Change in Time in Range (TIR) from inclusion to 12 months | Inclusion and 12 months
  Change in Time in Range (TIR, 70-180 mg/dL; for pregnant women: TIR, 63-140 mg/dL) (%), from inclusion (hybrid closed-loop initiation) to 12 months.
Change in Time In Tight Range (TITR) from inclusion to 3 months and 12 months | Inclusion, 3 and 12 months
  Change in Time In Tight Range (TITR, 70 - 140 mg/dL) (%) from inclusion (hybrid closed-loop initiation) to 3 months, and from inclusion to 12 months.
Change in Time Above Range (TAR) from inclusion to 3 months and 12 months | Inclusion, 3 months, and 12 months
  Change in Time Above Range (TAR, > 250 mg/dL and > 180 mg/dL; for pregnant women: TAR, > 140 mg/dL) (%) from inclusion (hybrid closed-loop initiation) to 3 months, and from inclusion to 12 months.
Change in Time Below Range (TBR) from inclusion to 3 months and 12 months | Inclusion, 3 and 12 months
  Change in Time Below Range (TBR, < 70 mg/dL and < 54 mg/dL; for pregnant women: TBR, < 63 mg/dL and < 54 mg/dL) (%) from inclusion (hybrid closed-loop initiation) to 3 months, and from inclusion to 12 months.
Change in average glucose levels from CGM sensor data from inclusion to 3 months, and to 12 months | Inclusion, 3 months and 12 months
  Change in average glucose levels from CGM sensor data (mg/dL) from inclusion (hybrid closed-loop initiation) to 3 months, and from inclusion to12 months.
Change in Standard Deviation (SD) of glucose from inclusion to 3 months, and to 12 months | Inclusion, 3 months and 12 months
  Change in Standard Deviation (SD) of glucose from sensor data from inclusion (hybrid closed-loop initiation) to 3 months, and from inclusion to 12 months
Change in Coefficient of Variation (CV) of glucose from inclusion to 3 months, and to 12 months | Inclusion, 3 months and 12 months
  Change in Coefficient of Variation (CV) of glucose derived from CGM sensor data (%) from inclusion (hybrid closed-loop initiation) to 3 months, and from inclusion to 12 months.
Change in Glucose Management Indicator (GMI) from inclusion to 3 months, and to 12 months | Inclusion, 3 months and 12 months
  Change in Glucose Management Indicator (GMI) (%) derived from CGM sensor data from inclusion (hybrid closed-loop initiation) to 3 months, and from inclusion to 12 months.
Change in HbA1c from inclusion to 3 months, and to 12 months | Inclusion, 3 months and 12 months
  Change in HbA1c (%) from inclusion (hybrid closed-loop initiation) to 3 months, and from inclusion to 12 months
Time in hybrid closed-loop | 3 months and 12 months
  Time spent in hybrid closed-loop (%) at 3 months and 12 months
System usage modalities at 3 months, and 12 months | 3 months and 12 months
  Description of evolution rate of advanced features (Boost mode and Ease-Off mode) at 3 months and 12 months, of the number of meal announcements per day, of the insulin-to-carbohydrate ratio, and alarms, at both 3 months and 12 months.
Change in the PAID questionnaire score from inclusion to 3 months, and to 12 months | Inclusion, 3 months and 12 months
  Self-administered questionnaire: Problem Areas In Diabetes (PAID)
  Following versions will be used: Adult version (18 and above), Teen version (PAID-T) in adolescents aged 12-18 years, and for their parents (P-PAID-T), Children version (PAID-C) in children aged 8-11 years and their parents (P-PAID-C). P-PAID-C will be also used in parents of children aged <8 years.
  The Problem Areas in Diabetes (PAID) questionnaire assesses diabetes-related emotional distress across patients and caregivers using age- and role-specific versions. The PAID (adults), PAID-T (teens), and PAID-C (children) are self-reported, while P-PAID-T and P-PAID-C are completed by parents of teens and children, respectively. All versions use Likert scales and are typically transformed to a 0-100 score, with higher values indicating greater distress.
  The PAID questionnaire will be completed at inclusion (hybrid closed-loop initiation), after 3 months and after 12 months.
Change in the DTSQ questionnaire score from inclusion to 3 months, and to12 months | Inclusion, 3 months and 12 months
  Self-administered questionnaire: Diabetes Treatment Satisfaction Questionnaire (DTSQs)
  Following versions will be used: Adult version (18 and above), Teen version (DTSQs-Teen) in adolescents aged 13-18 years. For their parents and parents of children aged <13 years, Parent version (DTSQs-Parent) will be used.
  DTSQQs for adults contains 8 items, DTSQs-Teen has 12 items and DTSQs-Parent has 14 items. The total score of the DTSQs is calculated by summing six items (excluding perceived hypo/hyperglycaemia), each rated 0 to 6, resulting in a total score from 0 to 36, with higher scores indicating better treatment satisfaction.
  The questionnaire will be completed at inclusion (hybrid closed-loop initiation), after 3 months and after 12 months.
Change in the HFS-II questionnaire score from inclusion to 3 months, and to 12 months | Inclusion, 3 months and 12 months
  Self-administered questionnaire Hypoglycemia Fear Survey II (HFS-II).
  The following versions will be used: Adult version, Children version (HFS-II children) for children aged 6 years and above, Parent version (HFS-II parent) for children aged 8 years and above, and Parent version for children aged <8 years (HFS-II parent of young children).
  HFS-II consists of items ranging from 0 (never) to 4 (almost always) (9 items in the Adult version, 25 in the Teen version and 26 in the Parent versions). It is composed of two subscales: a Behavior score and a Worry score, with higher scores reflecting greater behavioral or emotional impact.
  The questionnaire will be completed at inclusion (hybrid closed-loop initiation), after 3 months and after 12 months.
Change in the PSQI questionnaire score from inclusion to 3 months, and to 12 months | Inclusion, 3 months and 12 months
  Self-administered questionnaire: Pittsburgh Sleep Quality Index (PSQI).
  The questionnaire will be used in adults and parents. It contains 19 items which are grouped into 7 components that contribute to the overall score. Each component is scored from 0 to 3, where 0 indicates no difficulty and 3 indicates severe difficulty. The 7 component scores are summed to produce a total score ranging from 0 to 21.
  The questionnaire will be completed at inclusion (hybrid closed-loop initiation), after 3 months and after 12 months.
Perceived changes in quality of life, treatment satisfaction, fear of hypoglycemia, and sleep quality at 3 months, and at 12 months | Inclusion, at 3 months and 12 months
  Participant reported perceived changes in quality of life, treatment satisfaction, fear of hypoglycemia and sleep quality measured with a question " Patient Global Impression of Change " (PGIC) (one for each dimension) at 3 months, and at 12 months.
  Each PGIC will be used in adults, parents and children aged 11 years and above and consisting of one question with 7 modalities from 'Much worse" to "Much better".
Safety / Adverse events related to the use of the System | 3 months and 12 months
  The following events will be described at 3 months and 12 months: number of diabetic ketoacidosis events, severe hypoglycemia requiring assistance (medical and non-medical), diabetes-related work or school absences, unplanned hospitalizations related to diabetes and other complications related to the use of the system that meet the predefined acceptance criteria based on safety parameters for the target devices.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel SONNET, MD, Principal Investigator — Centre Hospitalier Universitaire de Brest - Cavale Blanche Hospital
Locations (20):
- France (20):
  - CHU Amiens, Amiens
  - Hôtel Dieu-Pédiatrie, Angers
  - CH Victor Dupouy, Argenteuil
  - Hôpital Bois Guillaume, Bois-Guillaume
  - CHU Brest - Hôpital La Cavale Blanche, Brest
  - Hôpital Femme Mère Enfant Lyon, Bron
  - CHU Grenoble Alpes, Grenoble
  - Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle
  - Hospices Civils de Lyon DIAB-Ecare, Lyon
  - Hôpital Européen, Marseille
  - Hôpital Europeen Georges Pompidou, Paris
  - Hôpital Universitaire Necker Enfants Malades, Paris
  - Groupe hospitalier Bichat Claude Bernard, Paris
  - CH Périgueux, Périgueux
  - CHU Poitiers, Poitiers
  - Hôpital NOVO, Site Pontoise, Pontoise
  - CHU Reims American Memorial Hospital, Reims
  - CHRU Nancy-Hôpitaux de Brabois Adultes, Vandœuvre-lès-Nancy
  - CH Bretagne Atlantique, Vannes
  - Hôpital Robert Schuman-UNEOS, Vantoux

IPD SHARING:
Plan to Share IPD: No
In accordance with the General Data Protection Regulation and French data protection laws the presentation of the results derived from data processing shall under no circumstances allow the direct or indirect identification of individuals participating in the study.
  In the event of publication of the study findings in a scientific journal, access to the data by an independent expert - including one appointed by a scientific publisher - shall only be granted through the interface provided or designated by the Data Controller, solely for the purpose of verifying or reproducing the analyses, and exclusively under the conditions defined for secure consultation and data handling. The study is a non-interventional trial.